CLINICAL TRIAL: NCT05573659
Title: Capillary Refill Time Calculated With a Video-assisted Method Has a Better Reproducibility Than Visual Method in Critically Ill Patients a Prospective Monocentric Study
Brief Title: Capillary Refill Time Calculated With a Video-assisted Method Has a Better Reproducibility Than Visual Method in Critically Ill Patients
Acronym: EVITREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0026
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Intensive Care Unit; Mortality; Reliability
Keywords: capillary refill time; intensive care unit; mortality; reliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video-assisted capillary refill time. (Experimental)
  Interventions: Other: video assisted cutaneous recoloration
- visual capillary refill time. (Active Comparator)
  Interventions: Other: time of cutaneous recoloration

INTERVENTIONS:
Other: time of cutaneous recoloration — In the shortest time possible (less than 3 minutes), realization of three successive measurements of the time of cutaneous recoloration by a pressure by the so-called visual method by two intensivists trained at the CRT of the surgical resuscitation service familiar with the technique of time of cutaneous recoloration. The measurements will be carried out blindly from each other.
  Arms: visual capillary refill time.
Other: video assisted cutaneous recoloration — Compression of the nail bed of the index of the subject studied until whitening of the pressed area, then release, the force will be equivalent to 300 g on a kitchen scale TPA 808S Techwood™ and time of compressions being of 5 seconds. Smartphone camera recording of the procedure (Iphone 7™, Apple Inc., Cupertino, CA). An assistant is in charge of timing the TRC between two "tops" given by the operator, the tops corresponding to the release of the pressure on the index so the beginning of the TRC and the total recoloration of the bleached area. This wizard records the three results in seconds with the associated tenth of a second.
  Arms: video-assisted capillary refill time.

SUMMARY:
Capillary refill time is the time it takes for the skin to regain its initial colour after moderate pressure. It is usually performed on the patient index finger, middle finger or ring finger with the examiner's thumb and index finger for five seconds, three measurements having to be averaged. Capillary refill time has a dependent operator character, but it has been shown to be accurately correlated with 14-day mortality in septic shock, hospitalisation need in pediatric population.

The purpose of this project is to show that capillary refill time obtained by a video-assisted method has a better inter- and intra-observer reproducibility than capillary refill time obtained by a visual method.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* hospitalized in ICU
* Patient or Family /relative with Inclusion Authorization

Exclusion Criteria:

* Pregnant or lactating women
* Under protection (guardianship, curators, reinforced curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Variation of measure of capillary refill time in visual assisted capillary refill time group. | 28 days
  Variation of capillary refill time measure between experimentors in visual assisted capillary refill time group.
Variation of measure of capillary refill time in video assisted capillary refill time group. | 28 days
  Variation of capillary refill time measure between experimentors in video assisted capillary refill time group.
Variation of measure of capillary refill time between both groups. | 28 days
  Variation of capillary refill time measure between experimentors between both groups

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No